CLINICAL TRIAL: NCT02820870
Title: Quality Improvement and Personalization for Statins (QUIPS) (QUE 15-286)
Brief Title: Quality Improvement and Personalization for Statins
Acronym: QUIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-002; QUE 15-286 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2016-05-23; First posted 2016-07-01 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Quality Improvement; Decision Support Tool; Performance Measurement; Primary Prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care Intervention Group (Experimental): Primary care providers will receive a generated print-out of statin recommendations for patient whose current medication therapy is not consistent with the new guidelines (i.e., are "guideline discordant"). Each day the research assistant will deliver a hardcopy of these patient specific recommendations to the teamlets for their use. In addition, providers will receive monthly audit and feedback reports on the percentage of their patients meeting the guidelines.
  Interventions: Behavioral: Statin Decision Support Intervention
- Usual Care Group (No Intervention): PACT teams that were not randomized to the intervention will serve as a usual care group and will be expected to follow the VA guidelines and HEDIS measures as part of the VA national roll-out.

INTERVENTIONS:
Behavioral: Statin Decision Support Intervention — The investigators have developed a "mock" medical record decision support tool for this project. Each week the investigators will pull a list of patients scheduled for a primary care visit at the Ann Arbor VAMC then calculate each patient's risk based on the clinical guidelines algorithm and compare the statin recommendation against their current prescriptions. For each patient whose current medication therapy is not consistent with the new guidelines (i.e., are "guideline discordant"), a brief recommendation will be generated. Each day the research assistant will deliver a hardcopy of these patient specific recommendations to the providers for their use. In addition, providers will receive monthly audit and feedback reports on the percentage of their patients meeting the guideline.
  Arms: Primary Care Intervention Group

SUMMARY:
The investigators developed novel quality improvement intervention consisting of a personalized decision support tool, an educational program, a performance measure, and an audit and feedback system to encourage the adoption of the VA/DoD guidelines for the use of statin medicines. The investigators then performed a cluster randomized trial of the intervention in a single clinic.

DETAILED DESCRIPTION:
The VA/DoD Committee on Clinical Practice Guidelines for the Management of Dyslipidemia for Cardiovascular Risk Reduction has created clinical practice guidelines that have been officially adopted by VA. The new guidelines are substantially different than previous guidelines, and arguably somewhat more complicated. Complicating matters somewhat, the American Heart Association and American College of Cardiology passed similar, but not identical, guidelines one year earlier and VA is also planning to adopt HEDIS (Healthcare Effectiveness Data and Information Set) performance measures for managing dyslipidemia, which are also similar, but not identical to the VA guidelines. Changing recommendations plus this misalignment - two guidelines, one performance measure, none identical or perfectly-understood - could create confusion and unclear guidance for practitioners.

The investigators are proposing a partnership with CAR and VA Ann Arbor Primary Care on a QI project to improve the adoption of these guidelines with a time and resource-efficient implementation strategy that will be tested in ten PACT teamlets.

As part of the larger project, the investigators have designed an efficient, multi-pronged intervention to improve statin use. The investigators first developed a preliminary intervention. The investigators then already conducted an assessment of the barriers and facilitators to implementation to obtain provider feedback to improve the planned intervention and develop ideas to make it better.

The intervention will have two parts. First, all clinicians at VA Ann Arbor received an educational session about the new guidelines. Second, the investigators have randomly divided the PACT teamlets in half. One half, "usual care," will receive all changes that VA in planning for the new guidelines.

The providers in the "intervention" group will receive the full intervention. This includes a personalized decision support tool for every guideline-discordant patient during the time of the intervention based on the VA guidelines. They will also receive automated personalized audit and feedback reports based on the guidelines that the investigators have developed together with VA's Center for Analytics and Reporting (CAR). Providers will also receive a poster in their clinical rooms alerting patients that the guidelines have changed.

Post-study clarification: The analysis divided the study in to three time periods. There was a period before the intervention (pre-QI) from December 12, 2015 to March 20, 2016; during the intervention (QI) from March 29-June 30, 2016, and after the intervention (post-QI) from July 1, 2016 to September 30, 2016. Each period was divided by study arm. All analyses were compared to the pre-QI baseline. Analyses were at the level of the patient visit. Eligible patients were those recommended statins by the VA/DoD clinical practice guidelines, but not receiving them.

ELIGIBILITY:
Inclusion Criteria: This was a clustered study. The investigators randomized five patient-aligned care teams (PACTS), intervened upon the physicians within each PACT, and evaluated the effect on individual patient visits.

* Eligible physicians were practicing PACT primary care physicians in the Ann Arbor VA Healthcare System.
* Eligible patients those who were seen in primary care during the period of analysis who were under 75 and who would be recommended a moderate-or-high-strength statin according to the VA/DoD guidelines, but were not on one at the time of the visit according to the electronic health record

Exclusion Criteria:

* Patient exclusion criteria included patients over the age of 75, or those who had an ICD-9 or ICD-10 codes for ESRD, muscle pain, pregnancy, or in-vitro fertilization in the 2 years prior to the study visit, those who were on moderate-or-high-strength statins, and those who were not eligible according to the guidelines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy B. Sussman, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Information security limitations would make it very difficult to share this data. Please contact the authors with any questions.

REFERENCES:
- [Derived] B Sussman J, Holleman RG, Youles B, Lowery JC. Quality Improvement and Personalization for Statins: the QUIPS Quality Improvement Randomized Trial of Veterans' Primary Care Statin Use. J Gen Intern Med. 2018 Dec;33(12):2132-2137. doi: 10.1007/s11606-018-4681-6. Epub 2018 Oct 3. PMID 30284172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All primary care providers at one VA Medical Center clinic were randomized prior to the start of the intervention. Eligible visits were those with patients who were recommended statins by VA/DoD guidelines, but were not receiving them. The intervention was only performed on intervention arm visits during the 3-month intervention duration.
Pre-assignment Details: The unit of analysis was the visit during the 3-month intervention, with clustering for provider. Patients who met VA/DoD statin recommendations were excluded from the project. Each time-period (pre-intervention, intervention, post-intervention) are visits, and hence should have different sample sizes.
Units Other Than Participants: Visits
Groups:
- Primary Care Intervention Group: Primary care providers received a personalized decision support tool, an educational program, and an audit and feedback system that evaluated appropriate patients. The intervention lasted 3 months. Providers results for the 3 months prior to the intervention and the 3 months after it ended were also analyzed as controls.
- Usual Care Group: PACT teams that were not randomized to the intervention also received the educational intervention, but otherwise engaged in usual care.
Period: Before Intervention
Arm/Group | Primary Care Intervention Group | Usual Care Group
Started (Care received prior to the intervention and intended to adjust for confounding due to chance.) | 15; 538 Visits (These are a separate set of visits from the intervention period and have different visit numbers.) | 28; 672 Visits (These are a separate set of visits from the intervention period and have different visit numbers.)
Completed | 15; 538 Visits | 28; 672 Visits
Not Completed | 0; 0 Visits | 0; 0 Visits
Period: Intervention
Arm/Group | Primary Care Intervention Group | Usual Care Group
Started | 15; 573 Visits | 28; 673 Visits
Completed | 15; 573 Visits | 28; 673 Visits
Not Completed | 0; 0 Visits | 0; 0 Visits
Period: Post Intervention
Arm/Group | Primary Care Intervention Group | Usual Care Group
Started (These are visits after the intervention was done. It tested the effects' persistence.) | 15; 603 Visits (These are a separate set of visits from the intervention period and have different visit numbers.) | 28; 728 Visits (These are a separate set of visits from the intervention period and have different visit numbers.)
Completed | 15; 603 Visits | 28; 728 Visits
Not Completed | 0; 0 Visits | 0; 0 Visits

BASELINE CHARACTERISTICS:
Population: These numbers reflect the number of primary care providers who were randomized to the Intervention Group and Usual Care Group.
Groups:
- Primary Care Intervention Group: Primary care providers will receive a generated print-out of statin recommendations for patient whose current medication therapy is not consistent with the new guidelines (i.e., are "guideline discordant"). Each day the research assistant will deliver a hardcopy of these patient specific recommendations to the teamlets for their use. In addition, providers will receive monthly audit and feedback reports on the percentage of their patients meeting the guidelines.
  Statin Decision Support Intervention: The investigators have developed a "mock" medical record decision support tool for this project. Each week the investigators will pull a list of patients scheduled for a primary care visit at the Ann Arbor VAMC then calculate each patient's risk based on the clinical guidelines algorithm and compare the statin recommendation against their current prescriptions.
- Total: Total of all reporting groups
Arm/Group | Primary Care Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 15 | 28 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (8.5) | 43.2 (8.1) | 44.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 5 | 15 | 20
Region of Enrollment [Number; unit: participants]
  United States | 15 | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percent of Visits Where Moderate-to-high-strength Statins Are Appropriately Initiated
Description: For a given visit during the study period for a patient who is guideline-appropriate for a moderate-to-high-strength statin but is not on one, the primary outcome is met if that patient is started on a moderate-or-high-strength statin within 30 days from the time of the visit, according to EHR medication data. The analysis was based on visits, not patients. It is possible that patients were included in more than one visit, as long as they were still guideline discordant.
Time Frame: 30 days
Population: Five care teams were randomized. Two with 15 total providers received the intervention. Three, with 28 providers, were the control arm. During the QI period, the intervention arm had 573 eligible visits and the control arm had 673. Our outcome was the chance an appropriate statin would be started at a visit.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Groups:
- Primary Care Intervention Group: Primary care providers will receive a generated print-out of statin recommendations for patient whose current medication therapy is not consistent with the new guidelines (i.e., are "guideline discordant"). Each day the research assistant will deliver a hardcopy of these patient specific recommendations to the teamlets for their use. In addition, providers will receive monthly audit and feedback reports on the percentage of their patients meeting the guidelines.
  Statin Decision Support Intervention: The investigators have developed a "mock" medical record decision support tool for this project. Each week the investigators will pull a list of patients scheduled for a primary care visit at the Ann Arbor VAMC then calculate each patient's risk based on the clinical guidelines algorithm and compare the statin recommendation against their current prescriptions. For each patient whose current medication therapy is not consistent with the new guidelines (i.e., are "guideline discordant"),
Arm/Group | Primary Care Intervention Group | Usual Care Group
Number analyzed (Participants) | 15 | 28
Number analyzed (Visits) | 573 | 673
Visits | 102 | 95
Statistical Analysis 1: Comparison: Primary Care Intervention Group vs Usual Care Group; Test type: Superiority; p < 0.01, Regression, Logistic; With clustering by provider and team; Odds Ratio (OR) = 3.00, 95% CI 2-sided [1.84 to 4.9]

2. Secondary Outcome: Percent of Visits in the Post-intervention 3 Months Where Moderate-to-high Strength Statins Are Appropriately Initiated
Description: To test the continued impact of the intervention, after the intervention was complete and both arms were receiving usual care we measured if a statin was started in the 30 days from the time of the visit among patients who are recommended moderate-to-high strength statins by the VA/DoD clinical practice guidelines, but were not on them at the time of their visit. This secondary outcome looks at the stability of the results after the intervention was stopped, not during the intervention. It is a different set of visits and has a different set of numbers from the intervention. During this period both groups received usual care.
Time Frame: 3 months
Population: Patient visits in the 3 months following the intervention with the same inclusion criteria used for the intervention. The analysis was based on visits, not patients. It is possible that patients were included in more than one visit, as long as they were still guideline discordant.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Primary Care Intervention Group | Usual Care Group
Number analyzed (Participants) | 15 | 28
Number analyzed (Visits) | 603 | 728
Visits | 57 | 95
Statistical Analysis 1: Comparison: Primary Care Intervention Group vs Usual Care Group; Test type: Superiority; p = 0.06, Regression, Logistic; With cluster by provider and team; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.99 to 2.77]

3. Secondary Outcome: Percent of Provider Response Forms Returned
Description: As a fidelity evaluation, the investigators will assess the rates at which providers return the provider response forms, which are given to understand why intervention providers did or did not alter care.
Time Frame: 3 months
Population: Whenever an intervention arm provider received a decision support reminder, they were also given a provider response form.
Measure: Count of Units; unit: Response forms
Units Other Than Participants: Response forms
Arm/Group | Primary Care Intervention Group
Number analyzed (Participants) | 15
Number analyzed (Response forms) | 573
Response forms | 211

4. Secondary Outcome: Responses on Provider Response Forms
Description: As a fidelity evaluation, the investigators will assess the reasons providers give for making or not making a clinical change during an intervention visit. We provided forms with check boxes for each of the outcomes listed.
Time Frame: 3 months
Population: Data represents the responses on the forms returned. The survey asked respondents if they made changes to their statins and to provide reasoning behind their decisions. Some selected more than one answer and some returned the survey that denoted yes/no but did not answer follow-up question elaborating on their decision.
Measure: Count of Units; unit: Response forms
Units Other Than Participants: Response forms
Arm/Group | Primary Care Intervention Group
Number analyzed (Participants) | 15
Number analyzed (Response forms) | 211
Response forms
  Provider changed statin prescription | 45
  Did not change due to: patient allergy | 26
  Did not change due to: no time during visit | 16
  Did not change due to: Already on statin | 25
  Did not change due to: status incorrect | 8
  Did not change due to: do not need statin | 8
  Did not change due to: patient refusal | 45

ADVERSE EVENTS:
Time Frame: The period during which adverse events could have occurred was 3 months.
Description: There were no adverse events.
Arm/Group | Primary Care Intervention Group | Usual Care Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/28
Other Adverse Events (participants affected / at risk) | 0/15 | 0/28

LIMITATIONS AND CAVEATS:
In our submitted publication we chose not to publish the fidelity evaluation, because we think it distracts from the findings of the paper.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes